CLINICAL TRIAL: NCT05671276
Title: Efficacy of Different Anti-Thrombotic Strategies on the Incidence of Silent Cerebral Embolism After Percutaneous Left Atrial Appendage Occlusion: a Randomized Control Trial
Brief Title: Efficacy of Different Anti-Thrombotic Strategies on the Incidence of Silent Cerebral Embolism After Percutaneous Left Atrial Appendage Occlusion
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Collaborators: Second Affiliated Hospital of Nantong University (Other); Jiangsu Taizhou People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-SR-228
Record Dates: First submitted 2023-01-03; First posted 2023-01-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Atrial Fibrillation; Left Atrial Appendage Occlusion; Silent Cerebral Embolism
Keywords: Atrial Fibrillation; Left Atrial Appendage Occlusion; Silent Cerebral Embolism; Oral Anticoagulation; Antiplatelet Therapy
MeSH Terms: conditions — Atrial Fibrillation | interventions — Aspirin; Clopidogrel; Rivaroxaban

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Antiplatelet Therapy (Active Comparator): DAPT (aspirin 100 mg and clopidogrel 75 mg) from 45 days to 6 month-follow-up, then aspirin alone
  Interventions: Drug: aspirin and clopidogrel
- Half-Dose NOAC (Experimental): Long-term half-dose NOAC (rivaroxaban 10 mg after 45 days)
  Interventions: Drug: Rivaroxaban

INTERVENTIONS:
Drug: aspirin and clopidogrel — DAPT (until 6 months) + ASA
  Arms: Standard Antiplatelet Therapy
Drug: Rivaroxaban — half-dose NOAC
  Arms: Half-Dose NOAC

SUMMARY:
The primary objective of this investigation is to compare the efficacy of two different antithrombotic strategies after percutaneous LAA occlusion with a Watchman device on the prevention of silent cerebral embolism.

DETAILED DESCRIPTION:
BACKGROUND Left atrial appendage intervention is increasingly recognized as an alternative strategy for thromboembolism prophylaxis in AF. Theoretically, a complete occlusion of left atrial appendage may eliminate the possibility of embolism from the appendage. However, residual risk exists due to blood stasis and endothelial dysfunction in the atrial fibrillation state. This may raise an issue that whether we should and how to give the patients after appendage occlusion long-term antithrombotic therapy.

Meanwhile, patients with AF have a high incidence of silent cerebral embolism (SCE), which has similar impact with clinical stroke on cognition function. We hypothesized that the SCE caused by micro embolism may act as part of the residual risk after appendage occlusion, thus, an optimal antithrombotic treatment to decrease the incidence of SCE remains unclear.

AIM OF THIS STUDY The primary objective of this investigation is to compare the efficacy of two different antithrombotic strategies after percutaneous LAA occlusion with a Watchman device on the prevention of SCE. The primary endpoint is incidence of SCE detected by MRI. The secondary endpoints are more than two new SCE detected by MRI, cognition function and composite endpoint of all-cause mortality, clinical thromboembolic events and major bleeding events.

DESIGN This is a randomized, prospective, multicenter design. We aim to include 150 patients 45 days after successful LAAC with WATCHMAN device. Patients are randomized in a 1:1 fashion into two arms: Standard Antiplatelet Therapy and Half-Dose NOAC. Follow-up duration of this study is 12 months. The 1-year routine follow-up strategy included DW-MRI scans performed approximately 90 days, 180 days, and 365 days post-procedure.

ELIGIBILITY:
Inclusion Criteria:

1. AF patients over 18 years old
2. Patients had undergone left atrial appendage occlusion with WATCHMAN device and confirmed no significant peri-device leak or DRT at the 45-day CT
3. Patients have a history of ischemic thromboembolic events or have CHA2DS2-VASc score ≥3

Exclusion Criteria:

1. Patients with an indication of long-term antiplatelet therapy other than LAAO at the time of enrollment (eg, ACS, Intracranial vascular stenosis≥75%)
2. Absolute contraindications to OAC
3. Absolute contraindications to anti-platelet therapy
4. Contraindications to MR or unwilling to receiving MR
5. Patients with clinical thromboembolicor major bleeding events within 45 days after LAA occlusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-09-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of silent cerebral embolism (SCE) detected by MRI | 45 days to 12 months
  New SCE at any MRI during the follow-up

SECONDARY OUTCOMES:
More than two new SCE detected by MRI | 45 days to 12 months
  More than two new SCE at any MRI during the follow-up, describing the number, location and the size.
Cognition function detected by MMSE test | 45 days to 12 months
  Cognition score detected by MMSE test
MoCA test | 45 days to 12 months
  Cognition score detected by MoCA test
Composite endpoint of of all-cause mortality, clinical thromboembolic events and major bleeding events | 45 days to 12 months
  Clinical thromboembolic including Ischemic stroke, Peripheral thromboembolic event, et al. Major bleeding including intracrania bleeding, gastrointestina bleeding et al.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided